CLINICAL TRIAL: NCT01759043
Title: Safety and Feasibility of Using a Single Transradial Guiding Catheter for Both Left and Right Coronary Angiography and Intervention in Patients With ST-segment Myocardial Infarction(RAPID)
Brief Title: Safety and Feasibility of Using a Single Transradial Guiding Catheter for Primary PCI
Acronym: RAPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Luhe Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-7071-01 CHRDS; CHRDS (Other Grant/Funding Number: The capital health research and development of sepcial)
Record Dates: First submitted 2012-12-24; First posted 2013-01-02 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Myocardial Infarction
Keywords: coronary artery disease; Myocardial Infarction; Radial Artery; Catheters
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- guiding catheter (Experimental): a single transradial guiding catheter for coronary angiography and intervention in patients with STEMI
  Interventions: Procedure: guiding catheter
- Diagnostic catheter (Active Comparator): Diagnostic catheter followed by guiding catheter selection for transradial primary PCI
  Interventions: Procedure: diagnostic catheter

INTERVENTIONS:
Procedure: guiding catheter — using a single transradial guiding catheter for coronary angiography and intervention
  Arms: guiding catheter
Procedure: diagnostic catheter — diagnostic for coronary angiography and guiding catheter selection for intervention
  Arms: Diagnostic catheter

SUMMARY:
The Rapid Trial is a randomized-controlled trial proposed to test the hypothesis that using a single guiding catheter for left and right coronary angiography and intervention in patients with ST elevation myocardial infarction (STEMI) can reduce procedure time, fluoroscopy time and Cath Lab door to balloon(C2B) time when compared with traditional approach which first underwent coronary angiography with diagnostic catheter followed by guiding catheter selection for intervention.

DETAILED DESCRIPTION:
1. background: Coronary intervention using transradial approach is common worldwide. It is normally necessary to use one diagnostic catheter and guiding catheter in primary percutaneous coronary intervention (PCI) for ST elevation myocardial infarction (STEMI). It is unknown whether using a single guiding catheter for both nonculprit and culprit vessel angiography and intervention during transradial primary percutaneous coronary intervention (PCI) is feasible.
2. objective:The aim of this study is to investigate the feasibility of using a single guiding catheter for left and right coronary angiography and intervention in patients with ST elevation myocardial infarction (STEMI).
3. This was a single-center, prospective, randomized study,patients with STEMI indicated for transradial primary PCI were randomized into two groups : group I consisted of patients who underwent coronary angiography and primary PCI by using a single guiding catheter.GroupII included patients who first underwent coronary angiography with diagnostic catheter followed by guiding catheter selection for intervention.
4. the primary Endpoints

   a.Cath Lab door to balloon time (C2B)
5. the Secondary endpoints:

   1. Occurrence of major adverse cardiac events (MACE) during 6 months

      * Cardiac death
      * Target vessel related myocardial infarction
      * Ischemia driven Target Vessel Revascularization (TVR)
      * Ischemia driven Target Lesion Revascularization (TLR)
      * Definite / probable stent thrombosis by ARC definition
   2. Number of catheters and wires used
   3. Vascular access complications (hematoma, aneurysm,pseudo-aneurysm, arteriovenous fistula formation, dissection, limb ischemia, bleeding)
   4. door to balloon time
   5. contrast consumption
   6. procedure time
   7. fluoroscopy time

ELIGIBILITY:
Inclusion Criteria:

* Patient must be > 18 years of age.
* Patients have typical chest pain for at least 20 minutes and have ECG changes typical for STEMI (ST elevation≥2mm in two continuous precordial leads or ST elevations≥1mm in two limb leads or new left bundle branch block) or ECG changes compatible with true posterior MI.
* Symptoms ≥ 30 min and ≤12 hours
* Patient and treating interventional cardiologist agree for randomization.
* Patient provides written informed consent.
* Diagnostic and therapeutic intervention performed through trans-radial/ulnar artery approach.
* Palpable radial or ulnar artery
* Previous experience of the operator with at least 100 cases of radial artery access within the past year

Exclusion Criteria:

* Concurrent participation in other investigational study
* Current platelet count <100 x 10^9cells/L or Hgb <10 g/dL.
* Absence of radial or ulnar artery pulsation
* Active bleeding or significant increased risk of bleeding, severe hepatic insufficiency, current peptic ulceration, proliferative diabetic retinopathy.
* Uncontrolled hypertension
* Prior CABG surgery
* Fibrinolytic therapy for current MI treatment
* patient have a life expectancy of <180days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cath Lab door to balloon time (C2B) | 24hours

SECONDARY OUTCOMES:
major adverse cardiac events (MACE) | 180days
  Cardiac death Target vessel related myocardial infarction Ischemia driven Target Vessel Revascularization (TVR) Ischemia driven Target Lesion Revascularization (TLR) Definite / probable stent thrombosis by ARC definition
Number of catheters and wires used | 24hours
Vascular access complications (hematoma, aneurysm,pseudo-aneurysm, arteriovenous fistula formation, dissection, limb ischemia, bleeding) | 30days
door to balloon time | 24hours
contrast consumption | 24hours
procedure time | 24hours
fluoroscopy time | 24hours

CONTACTS AND LOCATIONS:
Overall Officials: Jincheng Guo, M.D., Study Director — Beijing Luhe Hospital
Locations (1):
- Beijing Luhe hospital, Beijing, China

REFERENCES:
- [Result] Guo J, Chen W, Wang G, Liu Z, Hao M, Xu M, Zhu F. Safety and Efficacy of Using a Single Transradial MAC Guiding Catheter for Coronary Angiography and Intervention in Patients with ST Elevation Myocardial Infarction. J Interv Cardiol. 2017 Feb;30(1):33-42. doi: 10.1111/joic.12346. Epub 2016 Oct 25. PMID 27781297
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27781297/